CLINICAL TRIAL: NCT05979285
Title: Evaluation of Patient Experiences of Migraine Management and Feasibility of a Digital Headache Diary in Primary Care Setting: a Prospective Cohort Survey and Evaluative Study
Brief Title: MEDUSA Study - Migraine: Evaluation of Diagnosis, Utilisation of Services and Application
Acronym: MEDUSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumbria Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEDUSA1
Record Dates: First submitted 2023-07-14; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Migraine; Self-Assessment
Keywords: migraine; patient diary
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N1-Headache App (Experimental): All participants used the N1-HEadache App, a digital migraine diary that allows identification of triggers/protectors for migraine (as well as monitoring of medication use)
  Interventions: Device: N1-Headache App (by Curelator)

INTERVENTIONS:
Device: N1-Headache App (by Curelator) — Digital application allowing patients to monitor their migraines, and to identify triggers and/or protectors for their migraines.

SUMMARY:
Migraine is a very common condition characterised by frequent severe headaches that are very debilitating. Although the frequency and severity does reduce as patient's age, particularly above the age of 70, in younger and working age people this condition has a significant impact on people's lives. Patients with migraine are typically diagnosed and managed in primary care, but can also be treated by neurologists. Recently, NHS England has published guidance for clinical staff to optimise patient management: reduce admissions to hospital for migraine and improve the setting in which patients are seen. One recommendation is the increased use of headache diaries by patients. These may help patients and doctors to improve migraine diagnosis and its treatment, for example by identifying if there are triggers for getting a migraine attack. With technological advancements, there are now computer/phone applications (Apps) that can be used instead of a paper diary. The Curelator N1 Headache App is one of such migraine specific Apps. In this study, the investigators aim to evaluate if primary care migraine patients are open to using a digital headache diary App, and how compliant users of the App will be. The investigators also aim to assess patient feedback on the use of the N1 Headache App, and if its use aids them in the management of their migraine.

DETAILED DESCRIPTION:
Headaches are one of the most common ailments, and the headache disorder migraine is the second leading cause of years lived with disability. Some figures for the UK illustrate the extent of the issue: approximately 10 million people aged 15 - 69 live with migraine , and 3 million workdays are lost every year in to migraine-related absenteeism alone, at a cost of almost £4.4 billion. In the UK, the annual primary care consultation rate for headache is 4.4 per 100 registered patients, of whom 4% are referred to secondary care for further assessment. Headache and migraine is the top self-reported chronic condition amongst primary care patients. Management, including self-management, of migraine appears to be sub-optimal. Compliance with prophylactic therapy is poor with a limited number of patients using preventive treatment, even though many do try prophylactic medicines at some stage. After diagnosis there is often also a delay before preventive treatment is attempted, and commonly only tried once.

The issues related to migraine are worsening as reported by NHS England and in the national media : "NHS England has announced plans aimed at preventing up to 16,500 emergency hospital admissions for headaches and migraines each year. Greater use of headache diaries, where patients record their symptoms, and faster access to specialist advice for family doctors are among the measures intended to reduce the pressure on frontline services."

Headache diaries can be paper-based or electronic (Applications or Apps), and prospective or retrospective. Retrospective diaries are prone to under and overestimation by patients, and 'gaming' - completing e.g. a month worth of data at the end of that month - is a potential issue with prospective paper-based headache diaries. Electronic diaries may therefore offer a viable alternative to paper diaries. Numerous migraine diary Apps have been developed in the last decade, and some of them were found not user-friendly or did not measure clinically relevant outcomes. A more recent review on the topic of digital headache diaries concluded that patient and clinically relevant outcome measures for many were Apps were lacking. It is, however, recognised that headache diaries can aid patients and clinicians to track the course of a headache disorder, help to identify triggers and inform treatment plans. The usefulness of health Apps can be measured with a validated Mobile App Rating Scale.

Study aims and hypothesis

To assess if a digital headache diary App (Curelator N1 Headache) is an acceptable tool to monitor migraine in a cohort of primary care patients diagnosed with/coded for migraine by their GP practice. Furthermore, to determine the compliance rates achieved by users of the N1 Headache App.

ELIGIBILITY:
Inclusion Criteria:

* • Primary care patients diagnosed with or attending their GP practice ('coded for') migraine in the last 5 years. This may therefore be newly diagnosed patients or patients with long-standing migraine who attended their GP practice about their condition.

  * Patients aged ≥ 16 years
  * Mental capacity to give consent and not using an interpreter for GP consultations (ie competent in English and capacity to complete postal survey)
  * Part 2 only:

    * Completion of complete part 1 survey, including indication that patient still has ongoing migraine issues.
    * Access to email, internet and Apple or Android technology (ie smartphone, tablet or computer)

Exclusion Criteria:

* • Under the age of 16 years

  * Unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity
  * The patient has concurrent (medical) conditions that in the opinion of the investigator may compromise their capacity to complete the survey. Examples would be current severe ill health episode.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
patient interest in N1 Headache App | 30 days
  percentage of survey responders who indicate they are willing to trial the N1 Headache App
user compliance for N1 Headache App | 90 days
  percentage of participants who consent to using the App who comply with daily use in 90 day trial period

SECONDARY OUTCOMES:
previous use of digital diary Apps for migraine | 30 days
  what percentage of responders has previously used a digital diary App for migraine
usefulness of N1 Headache App: percentage patients who identify a migraine trigger | 90 days
  What percentage of patients who use the N1 Headache App often enough do identify a migraine trigger when a report is generated
Health Confidence and digital diary App | 90 days
  Does use of digital diary App for migraine affect patients' HEalth Confidence Score (Degree of agreeableness with statement 'I know enough about my migraine health', answers being 'disagree', 'neutral', 'agree' and 'strongly agree'

CONTACTS AND LOCATIONS:
Overall Officials: Stacey J Fisher, MD, Principal Investigator — substantive employee
Locations (1):
- Research & Development Department, Carlisle, Cumbria, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jonker L, Fitzgerald L, Vanderpol J, Fisher S. Digital diary App use for migraine in primary care: Prospective cohort study. Clin Neurol Neurosurg. 2022 May;216:107225. doi: 10.1016/j.clineuro.2022.107225. Epub 2022 Mar 25. PMID 35364371